CLINICAL TRIAL: NCT02855359
Title: An Open Label Phase 2 Study of Denintuzumab Mafodotin (SGN-CD19A) in Combination With RCHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone) or RCHP (Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone) Compared With RCHOP Alone as Frontline Therapy in Patients With Diffuse Large B-cell Lymphoma (DLBCL) or Follicular Lymphoma (FL) Grade 3b
Brief Title: Denintuzumab Mafodotin (SGN-CD19A) Combined With RCHOP or RCHP Versus RCHOP Alone in Diffuse Large B-Cell Lymphoma or Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN19A-004
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Diffuse, Large B-Cell, Lymphoma; Follicular Lymphoma, Grade 3b; Transformed Lymphoma / DLBCL
Keywords: Antibodies, Monoclonal; SGN-19A; Denintuzumab Mafodotin; DLBCL; Antibody-Drug Conjugate; Antigens, CD19; Hematologic Diseases; Immune System Diseases; Immunoproliferative Disorders; Immunotherapy; Lymphatic Diseases; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Monomethyl auristatin F; Neoplasms; Neoplasms by Histologic Type; Transformed Lymphoma / DLBCL; Cyclophosphamide; Doxorubicin; Liposomal doxorubicin; Prednisone; Rituximab; Vincristine; Alkylating Agents; Anti-Inflammatory Agents; Antibiotic, Antineoplastic; Antimitotic Agents; Antineoplastic Agents, Alkylating; Antineoplastic Agents; Phytogenic Antirheumatic Agents; Glucocorticoids; Drug Therapy; Follicular Lymphoma Grade 3b; immunosuppressive agents
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Hematologic Diseases; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Neoplasms; Neoplasms by Histologic Type | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- denintuzumab mafodotin + RCHOP (Experimental): Part A: denintuzumab mafodotin (SGN-CD19A) + RCHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone)
  Interventions: Drug: denintuzumab mafodotin; Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- denintuzumab mafodotin + RCHP (Experimental): Part A: denintuzumab mafodotin (SGN-CD19A) + RCHP (rituximab, cyclophosphamide, doxorubicin, and prednisone)
  Interventions: Drug: denintuzumab mafodotin; Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone
- denintuzumab mafodotin + RCHOP or RCHP (Experimental): Part B: denintuzumab mafodotin (SGN-CD19A) + RCHOP or RCHP
  Interventions: Drug: denintuzumab mafodotin; Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- RCHOP (Active Comparator): Part B: RCHOP alone: (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone)
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Drug: denintuzumab mafodotin — SGN-CD19A at 3 mg/kg will be administered every 6 weeks via intravenous (IV) infusion, up to a maximum of three (3) doses, on Day 1 of Cycles 1, 3, and 5 of 21-day cycles
  Arms: denintuzumab mafodotin + RCHOP; denintuzumab mafodotin + RCHOP or RCHP; denintuzumab mafodotin + RCHP
Drug: rituximab — 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Drug: cyclophosphamide — 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Drug: doxorubicin — 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Drug: vincristine — 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  Arms: RCHOP; denintuzumab mafodotin + RCHOP; denintuzumab mafodotin + RCHOP or RCHP
Drug: prednisone — 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles

SUMMARY:
This is a Phase 2 study to evaluate the combination of denintuzumab mafodotin in combination with RCHOP or RCHP compared with RCHOP alone as front-line therapy in patients with diffuse large B-cell lymphoma or follicular lymphoma Grade 3b.

DETAILED DESCRIPTION:
In Part A of the study, patients will be randomized 1:1 to receive denintuzumab mafodotin plus RCHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) or denintuzumab mafodotin plus RCHP (rituximab, cyclophosphamide, doxorubicin, and prednisone) to assess the safety of these 2 combination regimens. Part B of the study is designed to evaluate the antitumor activity and safety of denintuzumab mafodotin in combination with either RCHOP or RCHP (Experimental Arm) compared with RCHOP alone (Comparator Arm).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive patients with histologically confirmed systemic de novo or transformed diffuse large B-cell lymphoma (DLBCL) (from follicular or marginal zone lymphoma), or follicular lymphoma (FL) Grade 3b;

  * patients must have high intermediate or high risk disease
* Tumor tissue available from most recent biopsy to determine cell of origin
* Fluorodeoxyglucose-avid disease by positron emission tomography and measurable disease greater than 1.5cm diameter
* Eastern Cooperative Oncology Group performance status ≤2
* Age 18 years or older
* Adequate study baseline laboratory parameters

Exclusion Criteria:

* Previous history of treated indolent lymphoma
* History of another primary invasive cancer, hematologic malignancy, or myelodysplastic syndrome that has not been in remission for at least 3 years
* History of progressive multifocal leukoencephalopathy
* Cerebral/meningeal disease related to the underlying malignancy
* Patients with the following ocular conditions: corneal disorders, monocular vision (ie. best corrected visual acuity greater than or equal to 20/200 in one eye), or active ocular disorders requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pinelli, PA-C, MMSc., Study Director — Seagen Inc.
Locations (35):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Saint Bernards Cancer Center, Jonesboro, Arkansas
  - City of Hope, Duarte, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - University of Colorado Health Memorial Hospital, Colorado Springs, Colorado
  - Poudre Valley Hospital Harmony Campus, Fort Collins, Colorado
  - Central Georgia Cancer Care, Macon, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hattiesburg Clinic (Forrest General Hospital), Hattiesburg, Mississippi
  - Research Medical Center, Kansas City, Missouri
  - San Juan Oncology Associates, Farmington, New Mexico
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology / Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Health - Baylor University Medical Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Scott and White Memorial Hospital - Temple, Temple, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Vista Oncology INC PS, Olympia, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Ponce Medical School Foundation, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Started | 11 | 13 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 13 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0
Not completed — Study Termination by Sponsor | 9 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 80] | 72 [45 to 81] | 69 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0: Normal activity | 2 | 3 | 5
    1: Symptoms, but ambulatory | 8 | 5 | 13
    2: In bed less than 50% of the time | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part B Outcome Measure: Complete Response Rate (CR)
Description: Study did not progress to Part B.
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Part A and Part B Outcome Measure: Incidence of Adverse Events
Description: Part A data only; study did not progress to Part B.
Time Frame: 54.7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP
Number analyzed (Participants) | 11 | 13
Participants
  Any Treatment-emergent adverse event (TEAE) | 11 | 13
  Any Grade 3-5 TEAE | 11 | 12
  Any Treatment-related Adverse Event (AE) | 10 | 13
  Any DM treatment-related AE | 9 | 13
  Any RCHOP/RCHP treatment-related AE | 10 | 13
  Any AE with Outcome of Death | 2 | 1
  Any Serious Adverse Event (SAE) | 5 | 4
  Any Treatment-Related SAE | 4 | 3
  Any DM Treatment-Related SAE | 2 | 2

3. Primary Outcome: Part A and Part B Outcome Measure: Incidence of Laboratory Abnormalities
Description: Part A data reported; study did not progress to Part B. Laboratory abnormalities Grade 1+ are reported.
Time Frame: Up to 183 days
Measure: Count of Participants; unit: Participants
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP
Number analyzed (Participants) | 11 | 13
Participants
  Alanine aminotransferase increased | 3 | 4
  Hypoalbuminemia | 3 | 4
  Alkaline phosphatase increased | 5 | 8
  Aspartate aminotransferase increased | 5 | 9
  Blood bilirubin increased | 0 | 4
  Hypercalcemia | 3 | 0
  Hypocalcemia | 5 | 5
  Hyperglycemia | 8 | 11
  Hypoglycemia | 1 | 4
  Hypermagnesemia | 0 | 4
  Hypomagnesemia | 4 | 4
  Hypophosphatemia | 5 | 5
  Hypokalemia | 6 | 7
  Hypernatremia | 1 | 1
  Hyponatremia | 4 | 12
  Hyperuricemia | 0 | 1
  Anemia | 10 | 12
  Leukopenia | 10 | 13
  Lymphopenia | 9 | 13
  Neutropenia | 9 | 11
  Thrombocytopenia | 10 | 13

4. Secondary Outcome: Event-free Survival (EFS) Between Study Arms in Part B
Description: Study did not progress to Part B
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS) Between Study Arms in Part B
Description: Study did not progress to Part B.
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (OS) Between Study Arms in Part B
Description: Study did not progress to Part B.
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR) at End Of Treatment (EOT) Between Study Arms in Part B
Description: Study did not progress to Part B.
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Duration of Objective Response and of Complete Response (CR) Between Study Arms in Part B
Description: Study did not progress to Part B.
Time Frame: N/A - Endpoint not assessed
Population: Endpoint not assessed; study did not progress to Part B.
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP | Denintuzumab Mafodotin + RCHOP or RCHP | RCHOP
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 54.7 weeks
Arm/Group | Denintuzumab Mafodotin + RCHP | Denintuzumab Mafodotin + RCHOP
All-Cause Mortality (participants affected / at risk) | 2/11 | 2/13
Serious Adverse Events (participants affected / at risk) | 5/11 | 4/13
Other Adverse Events (participants affected / at risk) | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denintuzumab Mafodotin + RCHP (N=11) | Denintuzumab Mafodotin + RCHOP (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Hypotension (Vascular disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denintuzumab Mafodotin + RCHP (N=11) | Denintuzumab Mafodotin + RCHOP (N=13)
Vision blurred (Eye disorders) | 7 | 10
Neutropenia (Blood and lymphatic system disorders) | 6 | 8
Fatigue (General disorders) | 7 | 6
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Keratopathy (Eye disorders) | 5 | 6
Nausea (Gastrointestinal disorders) | 5 | 6
Dry eye (Eye disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Pyrexia (General disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Hypotension (Vascular disorders) | 2 | 4
Keratitis (Eye disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Headache (Nervous system disorders) | 4 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 3
Visual acuity reduced (Eye disorders) | 1 | 4
Asthenia (General disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Lacrimation increased (Eye disorders) | 1 | 3
Mucosal inflammation (General disorders) | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 3
Chills (General disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Eye pain (Eye disorders) | 2 | 1
Eye pruritus (Eye disorders) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Neutrophil count decreased (Investigations) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Photophobia (Eye disorders) | 1 | 2
White blood cell count decreased (Investigations) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Eye irritation (Eye disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Fungal infection (Infections and infestations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 2
Ocular toxicity (Eye disorders) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 2
Platelet count decreased (Investigations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Troponin increased (Investigations) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Asthenopia (Eye disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Corneal epithelium defect (Eye disorders) | 0 | 1
Corneal oedema (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Eye infection fungal (Infections and infestations) | 0 | 1
Eye oedema (Eye disorders) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was ended by sponsor prior to Part B enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT02855359/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT02855359/SAP_001.pdf